CLINICAL TRIAL: NCT00261001
Title: A Randomized Comparative Phase I Study to Evaluate and to Compare the Safety and Immunogenicity of a Transcutaneous Mode of Administration of a Licensed Tetanus/Influenza Vaccine to the Conventional Intramuscular Route of Vaccine Administration in Healthy Volunteers and HIV-infected Patients
Brief Title: Safety Study Comparing a Vaccine Transcutaneous Administration to the Intramuscular Route
Acronym: MANON-05
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Objectif Recherche Vaccins SIDA (Other)
Responsible Party: Pr Christine KATLAMA, Objectif Recherche Vaccins SIDA (ORVACS)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ORVACS 005
Record Dates: First submitted 2005-12-01; First posted 2005-12-02 (Estimated); Last update posted 2009-11-25 (Estimated); Status verified 2009-11

CONDITIONS: Healthy Volunteers; HIV Infection
Keywords: Transcutaneous; Vaccination; Safety; Immunogenicity; HIV; Treatment Experienced
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transcutaneous (Experimental)
  Interventions: Biological: Transcutaneous mode of administration
- Intramuscular (Active Comparator)
  Interventions: Biological: Intramuscular mode of administration

INTERVENTIONS:
Biological: Transcutaneous mode of administration
  Arms: Transcutaneous
Biological: Intramuscular mode of administration
  Arms: Intramuscular

SUMMARY:
The rationale for transcutaneous vaccination is based on the unique ability of cutaneous immune cells, especially Langerhans cells (LCs), to present antigens to the immune system. DCs can be found at high densities in the epidermis and the dermis of human skin, a fraction of which are the epidermal LCs. It is known that strong and efficient immune responses can be induced by targeting vaccines to skin APCs (Glenn 2003, Partidos 2003), e.g. by epicutaneous application of smallpox vaccine on scarified skin. Several obstacles however prevent vaccines from attaining sufficiently high and free concentrations in these target skin DCs.

In this clinical trial we aim at testing the safety and immunogenicity of this new transcutaneous route of vaccine administration, first with a licensed, well-known, safe and highly immunogenic vaccine i.e. Tetagrip® vaccine, which is licensed for subcutaneous (s.c.) and intra-muscular routes (i.m), and to compare the induced vaccine-specific immune responses to those induced with the conventional (i.m) injection. We hypothesize that the transcutaneous application of Tetagrip® in the commercially available standard preparation of 0.5 ml should be capable to induce at least similar antibody and CD4 and/or CD8 T cell responses to both the tetanus and the flu vaccinal antigens.

This Phase I, open label, randomized study is designed to evaluate and to compare the safety and immunogenicity of a transcutaneous mode of Tetanus / Influenza vaccination to the conventional i.m. route of vaccine administration in two cohorts: The cohort I constituted of healthy volunteers and the cohort II of HIV-infected patients in whom the virus is stably controlled by antiretroviral therapy, ensuring an immune competence and a capacity to respond to vaccines.

DETAILED DESCRIPTION:
The proposed study aims to translate our current knowledge about vaccinology, immunology of the skin and on transcutaneous penetration of epicutaneously applied active compounds, into the development of more efficient and well tolerated vaccines, and to progress toward an easy-to-apply patch system for transcutaneous application of vaccines.

To that purpose we aim at testing the safety and immunogenicity of a new transcutaneous route of vaccine administration. We propose to test this new route first with a well-known, safe and highly immunogenic vaccine i.e. anti-influenza and tetanus vaccine which is licensed for sub-cutaneous and intra-muscular routes, and to compare the vaccine-specific immune responses induced after transcutaneous administration to the conventional intramuscular (i.m) injection. Seasonal vaccination against influenza is recommended for all individuals at risk for severe flu, including persons above 60 years of age or suffering from chronic diseases and for medical personal. It is also highly recommended at any age to prevent influenza. In addition vaccination against tetanus is mandatory in childhood and requires recall injections every 5 years to protect against the lethal disease caused by the tetanus toxin.

We hypothesize that the transcutaneous application of a licensed anti-influenza-tetanus vaccine in the commercially available standard preparation of 0.5 ml should be capable to induce at least similar antibody and CD4 and/or CD8 T cell responses to both the tetanus and the flu vaccinal antigens.

Tetagrip® vaccine is an approved and commercially available vaccine manufactured by Sanofi-Pasteur, administered in one injection for preventive vaccination of adults against tetanus and influenza. The Tetagrip® vaccine therefore represents a safe and approved test vaccine to evaluate safety and immunogenicity of the mode of administration under investigation.

The long term goal of this strategy is to improve the efficacy of vaccines that are currently encountering major obstacles such as the HIV vaccines, and to develop a non invasive mode of vaccine administration. Results from this study will help establish a standardized study protocol for the application of HIV-vaccines in future clinical trials.

STUDY DESIGN This Phase I, open label, randomized on the vaccine administration route study is designed to evaluate and to compare the safety and immunogenicity of a transcutaneous mode of Tetanus / Influenza vaccination to the conventional i.m. route of vaccine administration in two cohorts: The cohort I constituted of healthy volunteers and the cohort II of HIV-infected patients in whom the virus is stably controlled by antiretroviral therapy, ensuring an immune competence and a capacity to respond to vaccines.

This is a multisite trial and is being conducted in Germany in two clinical centers:

Cohort I:

Charité - Universitätsmedizin Berlin Clinical Research Center for Hair and Skin Physiology Department of Dermatology and Allergy Schumannstr. 20/21 10117 Berlin, Germany.

Cohort II :

Hospital of the Johann Wolfgang Goethe-University Frankfurt am Main HIV Treatment & Research Unit Department of Internal Medicine II Theodor-Stern-Kai 7 60590 Frankfurt am Main -Germany

ELIGIBILITY:
Inclusion Criteria:

Cohort I

* Healthy male volunteers
* Negative HIV test within the last 3 months Cohort II
* HIV infected males
* Positive HIV-serology
* CD4+ counts > 350 cells/mm3 over the last year
* CD4 cells nadir >200/mm3
* Plasma HIV RNA < 400cp/ml over the last 6 months
* Efficient antiretroviral treatment with a minimum of three drugs since at least one year

In addition Patients from both cohorts must meet the following criteria to be eligible for the study:

* Age between 18 and 45 years,
* BMI between 21 - 26,
* Phototype I to IV
* Clinical examination and an interview on their medical history and possible current therapies
* Subjects able to receive vaccine administration by any of the two administration routes,
* Absence of tetanus vaccination within last 4 years,
* Absence of influenza vaccination in the last year,
* Absence of any psychological, familiar, sociological or geographical condition potentially hampering compliance with the study protocol schedule.
* Written informed consent

Exclusion Criteria:

In both cohorts, if any of the following apply, the subject cannot enter the study:

* Excessive terminal hair growth on the two investigational skin areas used for the transcutaneous mode of vaccination.
* Phototype V-VI
* Acute illness, e.g. fever, infection at screening and/or D0
* Any acute skin affection which may interfere with the trial assessment on the injection site,
* Any allergy or hypersensibility to one of the components of the Investigational Product (egg products, neomycin),
* Medical history of allergy or hypersensitization to any ingredient of colorant used in the transcutaneous mode of administration,
* Medical history of skin cancer,
* Any acute or chronic illness which may expose the subject or interfere with results of the trial,
* Use of any topical treatment on the injection site within the last four weeks,
* Use, within the past 3 months, of any topical and systemic treatment that would interfere with assessment and/or investigational treatment (anti-inflammatory drugs, immunosuppressors or any immune modulator agent),
* Prevision of UV sessions or sun exposure 6 weeks prior to the study or during the study period,
* Subjects with current alcohol or illicit drug use which, in the opinion of the investigator, may interfere with the subject's ability to comply with the dosing schedule and protocol evaluations.
* Subject being in the exclusion period of a previous clinical trial (1 month.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2005-10; Primary Completion 2006-02 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Clinical local and systemic tolerance to Tetagrip® vaccine administration for both transcutaneous (TC) and intramuscular (i.m) routes of administration .

SECONDARY OUTCOMES:
The protective tetanus and influenza-specific antibodies GMT titers.
The increase in tetanus and influenza specific antibody titers between baseline and day 14 and day 28.
The tetanus and influenza CD4 and CD8 peripheral blood T cells numbers.
The characteristics of vaccine-specific CD4 and CD8 T cell differentiation.
Proportion of responders with protective specific antibodies GMT titers

CONTACTS AND LOCATIONS:
Overall Officials: Christine Katlama, Professor/MD, Study Chair — Objectif Recherche Vaccin Sida; Ulrike Blume-Peytavi, Professor/MD, Principal Investigator — Charite University, Berlin, Germany; Brigitte Autran, Prof/MD/PhD, Study Chair — ORVACS
Locations (2):
- Germany (2):
  - Hospital of the Johann Wolfgang Goethe-University Frankfurt am Main, Frankfurt, Frankfurt Am Main
  - Charité - Universitätsmedizin Berlin, Berlin, State of Berlin

REFERENCES:
- [Background] Vogt A, Combadiere B, Hadam S, Stieler KM, Lademann J, Schaefer H, Autran B, Sterry W, Blume-Peytavi U. 40 nm, but not 750 or 1,500 nm, nanoparticles enter epidermal CD1a+ cells after transcutaneous application on human skin. J Invest Dermatol. 2006 Jun;126(6):1316-22. doi: 10.1038/sj.jid.5700226. PMID 16614727
- [Result] Vogt A, Mahe B, Costagliola D, Bonduelle O, Hadam S, Schaefer G, Schaefer H, Katlama C, Sterry W, Autran B, Blume-Peytavi U, Combadiere B. Transcutaneous anti-influenza vaccination promotes both CD4 and CD8 T cell immune responses in humans. J Immunol. 2008 Feb 1;180(3):1482-9. doi: 10.4049/jimmunol.180.3.1482. PMID 18209043
- [Derived] Combadiere B, Vogt A, Mahe B, Costagliola D, Hadam S, Bonduelle O, Sterry W, Staszewski S, Schaefer H, van der Werf S, Katlama C, Autran B, Blume-Peytavi U. Preferential amplification of CD8 effector-T cells after transcutaneous application of an inactivated influenza vaccine: a randomized phase I trial. PLoS One. 2010 May 26;5(5):e10818. doi: 10.1371/journal.pone.0010818. PMID 20520820